CLINICAL TRIAL: NCT07328594
Title: Impact of Daridorexant on Sleep, Daytime Alertness, and Smoking During Abstinence
Brief Title: Impact of Daridorexant on Sleep, Daytime Alertness, and Smoking
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Legacy Health System (Other)
Collaborators: Washington State University (Other)
Responsible Party: Principal Investigator, Barbara A. Sorg, Dow Neurobiology Chair, Legacy Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2233; 750140603 (Other Grant/Funding Number: Good Samaritan Foundation of Legacy Health)
Record Dates: First submitted 2025-12-30; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Smoking; Nicotine; Tobacco; Addiction; Substance Use Disorders; Insomnia; Sleep
Keywords: Insomnia; Daridorexant; Smoking; Nicotine; Tobacco; Sleep; Addiction; Substance use disorders
MeSH Terms: conditions — Smoking; Behavior, Addictive; Substance-Related Disorders; Sleep Initiation and Maintenance Disorders | interventions — daridorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Medical Monitor will remain blinded unless adverse event.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator)
  Interventions: Drug: Daridorexant 50 mg
- No treatment (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Daridorexant 50 mg — Active daridorexant vs placebo comparator in smokers with insomnia
  Arms: Treatment
Other: Placebo — Placebo in Smokers
  Arms: No treatment

SUMMARY:
Tobacco use is the leading cause of preventable death in the U.S., with 480,000 deaths per year and 7.7 million deaths globally. A major clinical symptom associated with abstinence from both licit and illicit drugs is insomnia, which is a clinically verified, major risk factor for relapse. Roughly half of the 40 million smokers in the U.S. attempt to quit annually, with very low rates of success. One major hurdle is poor sleep quality during abstinence. Compounding the problem is that some pharmaceuticals to help reduce smoking can increase insomnia. Poor sleep is recognized as a major impediment to maintaining abstinence from several drugs of abuse, including nicotine. Blockers of orexin have recently been proposed as a promising therapy for smoking cessation. Insomnia has been reported in up to 40% of smokers, and 80% report regular sleep disturbances, which can be amplified during abstinence. A new orexin blocker, daridorexant, was FDA approved within the past two years for the treatment of insomnia, and while it has been tested in healthy individuals with insomnia, it has not been tested in smokers, who suffer from insomnia, particularly during the withdrawal phase when trying to quit. Daridorexant has an improved profile of beneficial effects for those with insomnia, the most notable advantage being its shorter duration of action that promotes daytime alertness, which is problematic for both active smokers and smokers during withdrawal. Poor sleep leads to daytime sleepiness, which often leads to smoking to maintain alertness.

DETAILED DESCRIPTION:
The investigators will use a randomized, double-blind placebo-controlled design to determine how daridorexant given over 3 weeks of smoking abstinence will alter sleep, daytime alertness, and smoking behavior and craving for cigarettes. Sleep will be monitored using a sleep-tracking device, a sleep diary, and daytime alertness will be monitored using a performance metric (psychomotor vigilance task) three times per week for the 3 week study. Participants will also complete several other questionnaires related to smoking behaviors, craving, withdrawal, daytime sleepiness, and mood.

ELIGIBILITY:
INCLUSION

1. Adult participants who are cigarette smokers, 18-55 years of age.
2. Smokers: greater than 10 cigarettes/day.
3. Smoking for 1 year or longer.
4. Willingness to try to reduce or stay abstinent from cigarettes, smoking cessation aides (including nicotine gum or patches), smokeless tobacco, or electronic cigarettes for 3 weeks during the study.
5. Willingness to monitor sleep at home with an external device and maintain a simple sleep and smoking diary for 3 weeks.
6. Willingness to take a 5-min, mobile-based test 3X/day for 3 days/week during the 3 weeks.
7. Ability to travel to three Study Visits.
8. Are willing to abstain from consuming grapefruit products during the study.
9. Have an iPhone, best with iOS 17 or newer.

EXCLUSION:

1. Are currently taking any pharmaceutical drugs for smoking cessation, including: Nicotine patch or nicotine gum, buproprion (Wellbutrin, Zyban), varenicline (Chantix, Champix), other behavioral interventions such as cognitive behavioral therapy for smoking.
2. Are currently using cannabis or alcohol for sleep. Are currently taking any pharmaceutical drugs for insomnia, such as eszopiclone (Lunesta), zaleplon (Sonata) or zolpidem (Ambien, Ambien CR, Edluar, and Zolpimist) benzodiazepines, or opioids.
3. Are currently taking stimulants commonly used for ADHD, such as methylphenidate (Ritalin Concerta, Daytrana) or amphetamines (Adderall, Dexedrine, Vyvanse).
4. Are currently taking anti-seizure drugs, including lamotrigine, pregabalin (Lyrica), or gabapentin (Neurontin, Horizant, or Gralise).
5. Have non-nicotine substance dependence (diagnosed with substance use disorder, including alcohol or cannabis use disorder (current cannabis use is acceptable, and past illicit drug use is acceptable if greater than 2 months prior to testing and does not meet current criteria for substance use disorders (SUDs) according to DSM-5).
6. Have a major neurological disorder such as Parkinson's disease, epilepsy, Alzheimer's disease, multiple sclerosis, or any other serious neurological disorder.
7. Have a history of serious psychiatric disorders including bipolar disorder, schizophrenia, or suicidality.
8. Had a stroke or head injury which caused loss of consciousness for longer than three minutes in the past 1 year.
9. Are pregnant or breastfeeding.
10. Have been diagnosed with sleep apnea or other diagnosed sleep disorders such as narcolepsy.
11. Have been diagnosed with thyroid problems.
12. Have been diagnosed with COPD.
13. Have been doing variable shift work in the past 1 month or traveled more than 1 time zone in past month.
14. Are currently taking the following medications, supplements, or food: Daridorexant can interact with strong inhibitors of CYP3A4, which should be discussed with The Study Doctor's office (some of these include clarithromycin, diltiazem, erythromycin, itraconzale, ketoconazole, ritonavir, and verapamil).
15. Have a BMI of 33 or higher.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality | 2 days + 3 weeks study: 2 days to assess sleep prior to taking daridorexant followed by 3 weeks of daily daridorexant administration.
  Sleep device to assess: latency to sleep, number of awakenings during the night, and sleep stages.
Daytime alertness | Assessed 3 times per day (morning, midday, evening), 3 times per week for 3 weeks.
  Assess daytime alertness using a 5 min psychomotor vigilance task. Higher score indicates lower alertness.
Insomnia Severity Index | Assess at prescreening and on last day of the study (3 weeks and 2 days)
  Assesses extent of insomnia. Range is 0-28. Higher score indicates high level of insomnia.
Sleep Quality-sleep diary | Assessed 2 days prior to taking daridorexant and daily for 3 weeks during daily daridorexant administration.
  Daily sleep diary to assess self-reported sleep
Pittsburgh Sleep Quality Index | 2 days before beginning study medication.
  Assesses sleep quality (duration, disturbance, latency) over last 1 month. Range is 0-21; higher score indicates worse sleep quality.
PROMIS Sleep-Short Form 8a | 2 days before beginning study medication and last day of weeks 1, 2, 3.
  Assesses sleep quality over last 7 days. Range is 8-40, higher score indicates worse sleep/low alertness.
Karolinska Sleepiness Scale | Given 3X/day on days 3, 5, 7 of weeks 1, 2, 3.
  Assesses daytime alertness - single question. Range is 1-10. Higher score indicates lower alertness.

SECONDARY OUTCOMES:
Fagerstrom | Measure at pre-screening and at the end of each week for 3 weeks.
  Assesses extent of nicotine dependence. Range is 0-10. Higher score indicates higher dependence.
Smoking History and Habits | Measure at pre-screening.
  Must smoke 10 or more cigarettes per day.
Minnesota Scale Withdrawal from Nicotine | 2 days before beginning study medication, end of day on days 3, 5, 7 of weeks 1, 2, and 3.
  Assesses nicotine withdrawal symptoms over last 24 hr. Range is 0-60, higher score indicating higher withdrawal signs/symptoms.
QSU Brief Smoking Desire | End of day on days 3, 5, 7 of weeks 1, 2, and 3.
  Assesses desire to smoke. Range 7-49. Higher score indicates higher craving to smoke.
Number of cigarettes/vape products smoked | Reported daily for entire study (2 days + 3 weeks).
  Daily Sleep Diary includes number of cigarettes/vape products smoked.

OTHER OUTCOMES:
Morningness/Eveningness questionnaire | 2 days before beginning study medication
  Scores range from 16-83, with higher score indicating morning type and lower score evening type.
GAD-67 Anxiety | 2 days before beginning study medication and last day of the study (3 weeks, 2 days).
  Assesses anxiety levels over last 2 weeks. Range is 0-21, higher score indicating higher anxiety.
Patient Health Questionnaire 9 (PHQ 9 Depression) | 2 days before beginning study medication and last day of the study (3 weeks, 2 days).
  Assesses depression levels. Range is 1-27, higher score indicating higher depression.
Readiness to Quit | 2 days before beginning study medication and on last day of study (3 weeks, 2 days).
  Readiness to quit tobacco. Scale is 1-10, with higher score indicating more important to quit.

CONTACTS AND LOCATIONS:
Locations (1):
- Legacy Research Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mauries S, Rolland B, Mallevays M, Catoire S, Zehani F, Sauvage K, Davido G, Lejoyeux M, Geoffroy PA. Conditions of sleep restoration after smoking cessation: A systematic review. Sleep Med Rev. 2025 Apr;80:102041. doi: 10.1016/j.smrv.2024.102041. Epub 2024 Dec 9. PMID 39893864
- [Background] Ruuls SR, Sedgwick JD. Cytokine-directed therapies in multiple sclerosis and experimental autoimmune encephalomyelitis. Immunol Cell Biol. 1998 Feb;76(1):65-73. doi: 10.1046/j.1440-1711.1998.00715.x. PMID 9553778
- [Background] Fragale JE, James MH, Avila JA, Spaeth AM, Aurora RN, Langleben D, Aston-Jones G. The Insomnia-Addiction Positive Feedback Loop: Role of the Orexin System. Front Neurol Neurosci. 2021;45:117-127. doi: 10.1159/000514965. Epub 2021 May 28. PMID 34052815
- [Background] Hamidovic A. Dual Orexin Receptor Antagonists (DORAs) as an Adjunct Treatment for Smoking Cessation. CNS Drugs. 2022 May;36(5):411-417. doi: 10.1007/s40263-022-00918-0. Epub 2022 Apr 22. PMID 35451800
- [Background] Mignot E, Mayleben D, Fietze I, Leger D, Zammit G, Bassetti CLA, Pain S, Kinter DS, Roth T; investigators. Safety and efficacy of daridorexant in patients with insomnia disorder: results from two multicentre, randomised, double-blind, placebo-controlled, phase 3 trials. Lancet Neurol. 2022 Feb;21(2):125-139. doi: 10.1016/S1474-4422(21)00436-1. PMID 35065036